CLINICAL TRIAL: NCT04470193
Title: Self-management Intervention for Children With Chronic Medical Complexity: Pilot Feasibility Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: HRSA/Maternal and Child Health Bureau (U.S. Federal Agency)
Responsible Party: Principal Investigator, Flory Nkoy, Research Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 088596
Record Dates: First submitted 2020-07-06; First posted 2020-07-14 (Actual); Results first posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-07

CONDITIONS: Children With Medical Complexity
Keywords: medical complexity; multiple chronic conditions; children
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MyChildCMC Intervention Group (Experimental): Parents/patients randomized into the MyChildCMC Intervention Group will use the MyChildCMC app to monitor their child's daily symptoms for the duration of the study period (3 months). The MyChildCMC app includes a daily form consisting of 12 questions assessing child's vitals, pain, seizures, mood, and feeding as well as caregiver worry for the day. Daily reminders are sent to the parent to fill out the vitals form in the app. Parents/participants will also fill out a quality of life survey at baseline, 1 month, and 3 months as well as a caregiver satisfaction survey at 3 months.
  Interventions: Other: MyChildCMC app
- Standard of Care Group (No Intervention): Parents/patients randomized into the Standard of Care Group do not use the MyChildCMC app to monitor their child's daily symptoms and are instructed to continue with regular care for their child and to continue monitoring their child's symptoms on their own without the use of the app for the duration of the study period (3 months). Parents/participants will also fill out a quality of life survey at baseline, 1 month, and 3 months as well as a caregiver satisfaction survey at 3 months.

INTERVENTIONS:
Other: MyChildCMC app — Patients/parents will self-monitor their symptoms daily using the MyChildCMC app completing the daily vitals form. After patient/parents complete the daily form, the app provides in-app alerts and graphs showing symptom data over time.
  Arms: MyChildCMC Intervention Group

SUMMARY:
The investigators have developed a tool to facilitate self-management for children with medical complexity (complex, multisystem chronic diseases) called MyChildCMC (My Child's Complex Medical Condition). MyChildCMC is an online, phone application (app) that engages parents daily in ongoing monitoring of common, crosscutting acute symptoms, including respiratory distress, inadequate feeding/fluid intake, fever, altered mental status, pain, and seizure status. The MyChildCMC app also guides parents to recognize early warning signs for health deteriorations to avoid acute events (i.e., ED visits and/or hospitalizations).

Parent comments during the development of the MyChildCMC application revealed that the tool had potential in helping them manage their child's chronic conditions. This study will be the first to explore if online home monitoring using online technology is feasible, scalable, and can lead to improved CMC outcomes. This pilot trial for the MyChildCMC app was designed to determine preliminary impact by comparing outcomes (child QOL, child emergency department and hospital admissions, and parent/caregiver satisfaction with care) between the intervention and control groups. If successful, our approach will be a model for improving CMC care and reducing costs for families and children with medical complexity. Future MyChildCMC trials will integrate care coordination and a more robust alert system to help facilitate care and follow-up for patients.

DETAILED DESCRIPTION:
Aim: Investigators will assess the impact of the MyChildCMC app by comparing the following outcomes for the child and caregiver:

1. Child Quality of Life (QOL)
2. Child Emergency Department (ED) and hospital admissions
3. Number of hospital days
4. Parent/Caregiver satisfaction with care

ELIGIBILITY:
Participant Inclusion Criteria:

Children with complex medical conditions* ages 1 through 20 years with their primary caregiver (primary person caring for the child) who:

* have been seen at Primary Children's Hospital within 365 days,
* own a smartphone or a tablet computer with Internet access, and
* are English speaking *Physician diagnosis was used to determine CMC diagnosis

Exclusion Criteria:

* Critically ill children in imminent death
* Non-English speakers

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flory Nkoy, MD, MS, MPH, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kogan MD, Strickland BB, Newacheck PW. Building systems of care: findings from the National Survey of Children With Special Health Care Needs. Pediatrics. 2009 Dec;124 Suppl 4:S333-6. doi: 10.1542/peds.2009-1255B. No abstract available. PMID 19948596
- [Background] McPherson M, Arango P, Fox H, Lauver C, McManus M, Newacheck PW, Perrin JM, Shonkoff JP, Strickland B. A new definition of children with special health care needs. Pediatrics. 1998 Jul;102(1 Pt 1):137-40. doi: 10.1542/peds.102.1.137. No abstract available. PMID 9714637
- [Background] Newacheck PW, Strickland B, Shonkoff JP, Perrin JM, McPherson M, McManus M, Lauver C, Fox H, Arango P. An epidemiologic profile of children with special health care needs. Pediatrics. 1998 Jul;102(1 Pt 1):117-23. doi: 10.1542/peds.102.1.117. PMID 9651423
- [Background] Strickland B, McPherson M, Weissman G, van Dyck P, Huang ZJ, Newacheck P. Access to the medical home: results of the National Survey of Children with Special Health Care Needs. Pediatrics. 2004 May;113(5 Suppl):1485-92. PMID 15121916
- [Background] Cohen E, Berry JG, Camacho X, Anderson G, Wodchis W, Guttmann A. Patterns and costs of health care use of children with medical complexity. Pediatrics. 2012 Dec;130(6):e1463-70. doi: 10.1542/peds.2012-0175. Epub 2012 Nov 26. PMID 23184117
- [Background] Feudtner C, Villareale NL, Morray B, Sharp V, Hays RM, Neff JM. Technology-dependency among patients discharged from a children's hospital: a retrospective cohort study. BMC Pediatr. 2005 May 9;5(1):8. doi: 10.1186/1471-2431-5-8. PMID 15882452
- [Background] Dolk H, Parkes J, Hill N. Trends in the prevalence of cerebral palsy in Northern Ireland, 1981-1997. Dev Med Child Neurol. 2006 Jun;48(6):406-12; discussion 405. doi: 10.1017/S0012162206000909. PMID 16700928
- [Background] Farooqi A, Hagglof B, Sedin G, Gothefors L, Serenius F. Chronic conditions, functional limitations, and special health care needs in 10- to 12-year-old children born at 23 to 25 weeks' gestation in the 1990s: a Swedish national prospective follow-up study. Pediatrics. 2006 Nov;118(5):e1466-77. doi: 10.1542/peds.2006-1070. PMID 17079547
- [Background] Association CsH. Optimizing Health Care for Children with Medical Complexity Annual Report 2013:2.
- [Background] Vestal C. Improving Medicaid for 'Medically Complex' Kids. The Pew Charitable Trusts 2015;January 08.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was between June 2019 to December 2019. Recruitment occurred at Primary Children's Hospital in Salt Lake City, Utah.
Pre-assignment Details: Of the 68 subjects whose medical records were reviewed, 6 did NOT meet eligibility criteria (5 non-English speaking parents and 1 was on palliative care) and were NOT invited to participate. Of the 62 POTENTIALLY eligible subjects who were invited to participate in the study, 12 DECLINED to participate and WERE NOT enrolled, and 50 subjects AGREED to participate and were enrolled. Of the 50 subjects who were enrolled, 24 were randomized to MyChildCMC and 26 to usual care.
Period: Overall Study
Arm/Group | MyChildCMC Intervention Group | Standard of Care Group
Started | 24 | 26
Completed | 19 | 26
Not Completed | 5 | 0

BASELINE CHARACTERISTICS:
Population: Baseline population includes 50 participants (who AGREED to participate in the study and were enrolled ): 24 in the MyChildCMC group and 26 in the usual care group.
Groups:
- Usual Care Group: Parents/patients randomized into the Usual Care Group do not use the MyChildCMC app to monitor their child's daily symptoms and are instructed to continue with regular care for their child and to continue monitoring their child's symptoms on their own without the use of the app for the duration of the study period (3 months). Parents/participants will also fill out a quality of life survey at baseline, 1 month, and 3 months as well as a caregiver satisfaction survey at 3 months.
- Total: Total of all reporting groups
Arm/Group | MyChildCMC Intervention Group | Usual Care Group | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24 | 24 | 48
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 7.29 [1 to 17] | 9.65 [2 to 19] | 8.52 [1 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 15 | 14 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 20 | 18 | 38
  Hispanic | 3 | 8 | 11
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 24 | 26 | 50

OUTCOME MEASURES:

1. Primary Outcome: Patient Quality of Life (QOL)
Description: Compared Mean QOL Change from Baseline to Each Follow-up Assessment Between the Two study Groups, using the Ellzey et. al.'s QOL survey questionnaire for children with complex medical conditions, which assesses multiple domains including physical health, mental health, sleep, pain, activities and general QOL. The total QOL score was reported and standardized to 100 points, with scores ranging from 20 (the lowest QOL) to 100 (the highest QOL). Higher QOL scores represent a better outcome.
Time Frame: Quality of Life assessed at baseline, then compared to 1 month and 3 months from start of study/intervention
Population: Analysis included 50 participants at baseline (including 24 participants in the intervention group and 26 in the usual care group ), 40 participants at 1 months (including 16 in the intervention group and 24 in the usual care group), and 37 participants at 3 months (including 15 participants in the intervention and 22 participants in the usual care group).
Measure: Mean (Standard Deviation); unit: score on a scale, range from 20 to 100
Arm/Group | MyChildCMC Intervention Group | Usual Care Group
Number analyzed (Participants) | 24 | 26
score on a scale, range from 20 to 100
  Baseline QOL score | 62.7 (14.8) | 54.4 (15.0)
  1-month QOL score: number analyzed (Participants) | 16 | 24
  1-month QOL score | 59.8 (16.9) | 51.9 (12.2)
  3-month QOL score: number analyzed (Participants) | 15 | 22
  3-month QOL score | 55.2 (15.3) | 50.8 (15.6)
Statistical Analysis 1: Comparison: MyChildCMC Intervention Group vs Usual Care Group; We used a generalized estimating equation model for repeated assessments, with a common unstructured residual covariance matrix to account for correlation in repeated measurements in the same patient, to compare QoL total score at baseline, 1 month, and 3 months between the groups. We hypothesized that MyChildCMC users would have better outcomes for the child (higher QoL, fewer ED and/or hospital use and hospital days) and parent (higher satisfaction with child's care); Test type: Superiority — We approached 62 subjects to get a sample size of 50 participants, allowing up to 16% attrition, to estimate the proportions of patients satisfying dropout of 0.13 to within margins of error (half-widths of 90% Cis). The 50 evaluable subjects were used to estimate the SD of QoL, with a margin of error of ∼20%. The sample size also allowed us to provide provisional estimates of the effect size for the QoL outcome to within a margin of error of ±7.1 points, assuming a true SD of 15 points; p > 0.05, generalized estimating equation model

2. Secondary Outcome: Patient Emergency Department (ED)/Hospitalization
Description: Compare NUMBER of ED and hospital admissions 3-month pre, and 3-month post study initiation between the intervention and Usual care groups.
Time Frame: Change in ED/hospital admission between 3-month prior and 3-month post start of study/intervention
Population: Using intention-to-treat analysis, we compared numbers of ED/hospital admissions and hospital days (3-month pre- and 3-month post-enrollment; enrollment hospitalization excluded) between the groups using generalized linear models with logarithmic link and Poisson regression analysis, estimating rate ratios (RR) and 95% confidence intervals (CI). Covariates included age, sex, and race/ethnicity.
Measure: Mean (Standard Deviation); unit: number of ED and hospital admissions
Arm/Group | MyChildCMC Intervention Group | Usual Care Group
Number analyzed (Participants) | 24 | 26
number of ED and hospital admissions
  3-month pre-study | 1.13 (1.26) | 0.85 (1.05)
  3-month post-study | 1.08 (1.25) | 0.88 (1.11)
Statistical Analysis 1: Comparison: MyChildCMC Intervention Group vs Usual Care Group; Test type: Superiority; p = 0.882, Mixed Models Analysis; Risk Ratio (RR) = 1.05, 95% CI 2-sided [0.58 to 1.88]

3. Secondary Outcome: Number of Hospital Days
Description: Number of days (duration) participants were hospitalized
Time Frame: 3-month pre and 3-month post study start
Population: Number of hospital days were compared between the Intervention group participants and Usual Care group participants.
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Intervention Group: Participants randomized to MyChildCMC intervention
- Usual Care Group: Participants randomized to continue with their usual care
Arm/Group | Intervention Group | Usual Care Group
Number analyzed (Participants) | 24 | 26
Days
  3-Month Pre | 9.25 (18.30) | 1.08 (1.88)
  3-Month Post | 4.54 (6.95) | 2.46 (3.84)
Statistical Analysis 1: Comparison: Intervention Group vs Usual Care Group; Test type: Superiority; p < 0.001, Mixed Models Analysis; Risk Ratio (RR) = 0.49, 95% CI 2-sided [0.39 to 0.62]

4. Secondary Outcome: Parent/Caregiver Satisfaction With Care
Description: Caregiver satisfaction with overall care of their children, using an adapted version (by Ellzey et. al) of Client Satisfaction Questionnaire for children with complex medical conditions, which has 6 questions measuring caregiver's confidence with ability to take care of child's health, consistency in doing things needed to take care of the child, availability of medical professional support, availability of social support, availability of a monitory system to help with child's home care and stress about child's health. We reported the total caregiver satisfaction scores, which range from 5 (the lowest satisfaction) to 30 (the highest satisfaction). Higher caregiver satisfaction scores represent a better outcome.
Time Frame: Collected once at study end (3 months)
Measure: Mean (Standard Deviation); unit: score on a scale, ranging from 5 to 30
Arm/Group | MyChildCMC Intervention Group | Usual Care Group
Number analyzed (Participants) | 24 | 26
score on a scale, ranging from 5 to 30 | 26.93 (2.22) | 24.14 (4.21)
Statistical Analysis 1: Comparison: MyChildCMC Intervention Group vs Usual Care Group; Test type: Superiority; p = 0.035, Mixed Models Analysis; Risk Ratio (RR) = 1.11, 95% CI 2-sided [1.01 to 1.22]

ADVERSE EVENTS:
Time Frame: The study lasted 3 months and adverse events were collected during the study 3-month period
Description: This was a minimal risk study and there was no adverse event related to the intervention during the study period.
Groups:
- Usual Care Group: Parents/patients randomized into the Standard of Care Group do not use the MyChildCMC app to monitor their child's daily symptoms and are instructed to continue with regular care for their child and to continue monitoring their child's symptoms on their own without the use of the app for the duration of the study period (3 months). Parents/participants will also fill out a quality of life survey at baseline, 1 month, and 3 months as well as a caregiver satisfaction survey at 3 months.
Arm/Group | MyChildCMC Intervention Group | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 2/24 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 0/24 | 0/26

LIMITATIONS AND CAVEATS:
Baseline hospital days were imbalance, due to small sample size and data skewing. Analysis accounted for skewness and baseline number of ED/hospital admissions were similar, minimizing allocation bias. We had 2 deaths and 1 hospice discharge in MyChildCMC group, suggesting sicker subjects in this group due to our small sample size, or despite sicker children in MyChildCMC group, hospital days dropped but increased in controls, suggesting the effect size may be larger.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-12): https://cdn.clinicaltrials.gov/large-docs/93/NCT04470193/Prot_SAP_000.pdf